CLINICAL TRIAL: NCT00357214
Title: Effect of Potassium Bicarbonate on Bone and Muscle
Brief Title: Effect of Potassium Bicarbonate Supplementation on Bone and Muscle in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Bess Dawson-Hughes, Senior Scientist, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01AR052322 (NIH); R01AR052322 (NIH)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Osteoporosis; Sarcopenia
Keywords: bone turnover; calcium excretion; nitrogen excretion; potassium bicarbonate; muscle loss; muscle atrophy; bone loss
MeSH Terms: conditions — Osteoporosis; Sarcopenia; Muscular Atrophy; Bone Diseases, Metabolic | interventions — potassium bicarbonate; Sodium Bicarbonate; Potassium Chloride; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- potassium bicarbonate (Active Comparator): Participants will receive potassium bicarbonate in dosage of 67.5 mmol/d. This compound has no other name.
  Interventions: Dietary Supplement: Potassium Bicarbonate
- Sodium bicarbonate (Active Comparator): Participants will receive sodium bicarbonate in dosage of 67.5 mmol/d. This compound has no other name.
  Interventions: Dietary Supplement: Sodium Bicarbonate
- Potassium chloride (Active Comparator): Participants will receive potassium chloride in dosage of 67.5 mmol/d. This compound has no other name.
  Interventions: Dietary Supplement: Potassium Chloride
- microcrystalline cellulose (Placebo Comparator): Participants will receive placebo is microcrystalline cellulose. This compound has no other name.
  Interventions: Dietary Supplement: placebo (microcrystalline cellulose)

INTERVENTIONS:
Dietary Supplement: Potassium Bicarbonate — 67.5 mmol/d given as three tablets after each meal, with a full glass of water
  Arms: potassium bicarbonate
Dietary Supplement: Sodium Bicarbonate — 67.5 mmol/d given as three tablets after each meal, with a full glass of water
  Arms: Sodium bicarbonate
Dietary Supplement: Potassium Chloride — 67.5 mmol/d given as three tablets after each meal, with a full glass of water
  Arms: Potassium chloride
Dietary Supplement: placebo (microcrystalline cellulose) — Given as three tablets after each meal, with a full glass of water
  Arms: microcrystalline cellulose

SUMMARY:
There is increasing evidence that the acid-base balance of diet plays an important role in the health of bones and muscles. An excess of acid in the body can result in calcium loss and muscle breakdown. Potassium bicarbonate, a base supplement, can neutralize acid within the body. The purpose of this study is to determine the effectiveness of potassium and bicarbonate, alone and combined, at reducing bone loss and preventing muscle wasting in older adults.

DETAILED DESCRIPTION:
The typical American diet of dairy products, grains, and meats results in excess acid build-up in the body. The kidney is often unable to remove this excess acid quickly enough, resulting in mildly elevated blood acidity. In an attempt to neutralize the acidity, the body releases calcium from its bones. Over time, however, this calcium loss can lead to decreased bone density and possibly osteoporosis. Excess acid in the body also stimulates the breakdown of muscle. The combination of osteoporosis and reduced muscle strength sets the stage for falls, fractures, and ultimately functional decline. At least 30% of older adults fall once a year and, of those falls, 5% result in fractures. Preserving muscle mass and strength is an effective way to lower the risk of falling and to maintain independence among older people. Potassium bicarbonate is a base supplement that can neutralize acid. The purpose of this study is to determine the effectiveness of potassium and bicarbonate, alone and combined, at reducing bone loss and preventing muscle wasting in older adults.

This study will last 3 months. Participants will be randomly assigned to one of four treatment groups:

* Group 1 will receive potassium bicarbonate supplements
* Group 2 will receive potassium chloride supplements
* Group 3 will receive sodium bicarbonate supplements
* Group 4 will receive placebo supplements

All participants will take three pills of their assigned supplement after each meal; this will occur on a daily basis throughout the study. Participants will also take a multivitamin and a 600-mg calcium tablet daily. Participants will not be required to alter their usual diet in any way, but they will be requested to not take their usual calcium and vitamin D supplements during the study. Study visits will occur on Days 1, 21, 49, and 84. Days 1 and 84 study visits will include a review of medical history and physical activity, blood collection, and evaluation of weight, blood pressure, calcium absorption, and muscle function. Collection of both a 24-hour urine sample and a calendar depicting compliance with the supplement schedule will also occur at these two visits. The other study visits, on Days 21 and 49, may include blood collection, calendar compliance checking, and weight and blood pressure measurements. Supplements will be handed out on Days 1, 21, and 49.

ELIGIBILITY:
Inclusion Criteria:

* Body mass idex less than 35
* Not currently on a weight gain or weight loss diet
* Willing to maintain usual level of physical activity
* Willing to refrain from taking own calcium supplements, antacids, or salt substitutes

Exclusion Criteria:

* Vegetarian
* Use of glucocorticoids for more than 10 days in the 3 months prior to study entry
* Use of estrogen, raloxifene, or calcitonin in the 6 months prior to study entry
* Use of bisphosphonate or teriparatide in the 2 years prior to study entry
* Current use of diuretics, nonsteroidal anti-inflammatory drugs (NSAIDS), beta-blockers, anabolic drugs (steroids or other), angiotensin converting enzyme (ACE) inhibitors, or angiotensin receptor blockers (ARBs)
* Renal disease, including kidney stones in the 5 years prior to study entry or creatinine clearance less than 50 ml/min/1.73 m2 of body surface area
* Hyperparathyroidism
* Untreated thyroid disease
* Significant immune disorder
* Current unstable heart disease
* Active malignancy or cancer therapy in the year prior to study entry
* 24-hour urine calcium levels greater than 300 mg/d after 1 week of being off calcium supplements
* Hypertension, congestive heart failure, arrythmias, or myocardial infarction in the 12 months prior to study entry
* On a salt-restricted diet
* Bone density total hip T score of less than -2.5
* Abnormal serum calcium
* Alkaline phosphatase levels greater than 10% above the upper end of the reference range
* Adrenal insufficiency, primary aldosteronism, or Bartter's syndrome
* Diabetes mellitus
* Alcohol use exceeding two drinks/day
* Peptic ulcers or esophageal stricture
* Screening serum 25(OH)D levels below 16 ng/ml

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bess Dawson-Hughes, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Result] Dawson-Hughes B, Harris SS, Palermo NJ, Castaneda-Sceppa C, Rasmussen HM, Dallal GE. Treatment with potassium bicarbonate lowers calcium excretion and bone resorption in older men and women. J Clin Endocrinol Metab. 2009 Jan;94(1):96-102. doi: 10.1210/jc.2008-1662. Epub 2008 Oct 21. PMID 18940881
- [Result] Dawson-Hughes B, Castaneda-Sceppa C, Harris SS, Palermo NJ, Cloutier G, Ceglia L, Dallal GE. Impact of supplementation with bicarbonate on lower-extremity muscle performance in older men and women. Osteoporos Int. 2010 Jul;21(7):1171-9. doi: 10.1007/s00198-009-1049-0. Epub 2009 Sep 1. PMID 19727904
- [Derived] Harris SS, Dawson-Hughes B. No effect of bicarbonate treatment on insulin sensitivity and glucose control in non-diabetic older adults. Endocrine. 2010 Oct;38(2):221-6. doi: 10.1007/s12020-010-9377-6. Epub 2010 Jul 17. PMID 21046483

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Potassium Bicarbonate | Sodium Bicarbonate | Potassium Chloride | Microcrystalline Cellulose
Started | 43 | 43 | 42 | 43
Completed | 39 | 39 | 42 | 42
Not Completed | 4 | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Potassium Bicarbonate | Sodium Bicarbonate | Potassium Chloride | Microcrystalline Cellulose | Total
Number analyzed (Participants) | 43 | 43 | 42 | 43 | 171
Age, Customized [Mean (Standard Deviation); unit: years]
  participant age | 62.2 (7.6) | 62.6 (7.6) | 63.4 (7.7) | 63.3 (7.7) | 62.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 24 | 25 | 97
  Male | 19 | 19 | 18 | 18 | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 43 | 43 | 42 | 43 | 171

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Markers of Bone Turnover
Description: Change in 24-hr urinary N-telopeptide/creatinine measured at baseline and 3 months
Time Frame: 3 month change in 24-hr urine values
Measure: Mean (Standard Error); unit: nmol/mmol
Arm/Group | Potassium Bicarbonate | Sodium Bicarbonate | Potassium Chloride | Microcrystalline Cellulose
Number analyzed (Participants) | 39 | 39 | 42 | 42
nmol/mmol | -6.25 (1.75) | -3.36 (1.68) | -0.14 (1.71) | 0.5 (1.61)

ADVERSE EVENTS:
Arm/Group | Potassium Bicarbonate | Sodium Bicarbonate | Potassium Chloride | Microcrystalline Cellulose
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 1/43 | 3/43 | 7/42 | 1/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Potassium Bicarbonate (N=43) | Sodium Bicarbonate (N=43) | Potassium Chloride (N=42) | Microcrystalline Cellulose (N=43)
gastrointestinal symptoms (Gastrointestinal disorders) | 1 (1) | 3 (3) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No